CLINICAL TRIAL: NCT00962195
Title: The Effect of Purple Sweet Potato (PSP)-Juice on Liver Enzymes and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: E. Boelsma, PhD, TNO Quality of Life, Business unit biosciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P8604
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: Health; Blood Pressure; Liver Function; Insulin Resistance
Keywords: health; blood pressure; liver enzymes; insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- purple sweet potato juice (Experimental): Daily oral intake of 3x 125 ml of PSP-juice for a period of 8 weeks
  Interventions: Dietary Supplement: purple sweet potato (PSP)-juice
- Control juice (Placebo Comparator): Daily oral intake of 3x 125 ml of control juice for a period of 8 weeks
  Interventions: Dietary Supplement: purple sweet potato (PSP)-juice

INTERVENTIONS:
Dietary Supplement: purple sweet potato (PSP)-juice — Daily oral intake of 3x 125 ml of PSP-juice or control juice

SUMMARY:
Purple Sweet Potato juice (PSP-juice) is a juice based on purple-fleshed sweet potato concentrate, containing a high level of anthocyanins. Purple-fleshed sweet potatoes have attracted attention to industry and scientists due to multiple physiological functions such as radical-scavenging, ACE-inhibitory and α-glucosidase inhibitory activities in vitro, and also hepato-protective, antihypertensive and antihyperglycemic effects in vivo. Previous studies in Japanese subjects showed potential beneficial effects of PSP beverages on liver function and blood pressure in volunteers with impaired hepatic function and/or hypertension.

The main objective of this study is to examine the effect of PSP-juice on liver enzymes and blood pressure. The secondary objective is to examine the effects of PSP-juice juice on insulin resistance.

DETAILED DESCRIPTION:
Study design: The study is designed as a randomized, parallel, placebo-controlled, double-blind study.

Study population: 40 healthy adult female and/or male subjects, 40-70 yr old with a BMI 25-35 kg/m2, mildly elevated serum liver enzymes, and high normal blood pressure or mild hypertension.

Intervention: Daily oral intake of 3x 125 ml of PSP-juice or control juice for a period of 8 weeks.

Main study parameters/endpoints: Liver enzymes (GGT, ALAT, ASAT), blood pressure, glucose, insulin, haematology and serum clinical chemical profile

ELIGIBILITY:
Inclusion Criteria:

* Healthy as assessed by the: Health and Lifestyle Questionnaire, results of the pre study laboratory tests in blood
* Males/Females aged 40-70 years (boundaries included) at Day 01 of the study
* Body Mass Index (BMI) 25-35 (boundaries included) kg/m2
* Liver enzymes above reference values GGT ≥ 45 IU/L (for males) and ≥ 35 IU/L (for females), and/or ASAT ≥ 45 IU/L (for males and females), and/or ALAT ≥ 50 IU/L (for males) and ≥ 40 IU/L (for females)
* Blood pressure (automated measurements at site): systolic blood pressure 130-159 mm Hg (boundaries included) and/or diastolic blood pressure 85-99 mm Hg (boundaries included)
* Voluntary participation
* Having given written informed consent
* Willing to comply with the study procedures
* Willing to give up blood/plasma donation during the study
* Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
* Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
* Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances
* Having a history of medical or surgical events that may significantly affect the study outcome
* Any concomitant medication, with the exception of occasional use of a paracetamol tablet, that may influence the outcome of the study (to be judged by the medical investigator)
* Food allergy/intolerance
* Alcohol consumption > 28 units/week for males and > 21 units/week for females
* Smoking > 10 cigarettes per day
* Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre study screening
* Reported slimming or medically prescribed diet
* Participation in night shift work
* Pregnant or lactating or wishing to become pregnant in the period of the study
* Personnel of TNO Quality of Life, their partner and their first and second degree relatives
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding his/her health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
liver enzymes | every 2 weeks during 8-weeks intervention

SECONDARY OUTCOMES:
blood pressure | every 2 weeks during 8-weeks intervention
insulin resistance | every 2 weeks during 8-weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Esther Boelsma, PhD, Principal Investigator — TNO; Ineke Klopping-Ketelaars, PhD, Study Director — TNO
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands